CLINICAL TRIAL: NCT01066676
Title: Prospective, Clinical Trial to Investigate Safety, Tolerability and Efficacy of Dexibuprofen Gebro 400 mg Powder for Oral Suspension (Test) Compared to Ibuprofen 400 mg Powder for Oral Suspension (Reference) in Patients Suffering From Osteoarthritis of the Hip or Knee
Brief Title: Dexibuprofen 400 mg Sachet Versus Ibuprofen 400 mg Sachet in Patients With Osteoarthritis of the Hip or Knee
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gebro Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IV/48.4
Record Dates: First submitted 2010-02-09; First posted 2010-02-10 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Osteoarthritis of the Hip or Knee
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — dexibuprofen; Ibuprofen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexibuprofen (Experimental): Dexibuprofen 400 mg powder for oral suspension
  Interventions: Drug: Dexibuprofen
- Ibuprofen (Active Comparator): Ibuprofen 400 mg powder for oral suspension
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Dexibuprofen — 400mg powder for oral suspension, daily dose 800mg
  Arms: Dexibuprofen
Drug: Ibuprofen — 400mg, powder for oral suspension, daily dose 1600mg
  Arms: Ibuprofen

SUMMARY:
Medical condition under investigation: Osteoarthritis of the hip or knee

Number of patients planned: 480 adult patients

Main objective: To evaluate and compare the tolerability profile of Dexibuprofen Gebro 400 mg powder for oral suspension compared to Ibuprofen 400 mg in patients with painful osteoarthritis of the hip or knee

Secondary objectives: To compare the overall efficacy of Dexibuprofen Gebro 400 mg powder for oral suspension compared to Ibuprofen 400 mg in patients suffering from different complaints due to painful osteoarthritis of the hip or knee

ELIGIBILITY:
Inclusion Criteria:

* male or female patients aged between 18 and 75 years
* everyday joint pain for the past three months
* global pain intensity in the involved joint (hip or knee) of "moderate" to "severe" within the last 48 h

Exclusion Criteria:

* acute inflammation or ischaemic necrosis
* paget's disease, chondrocalcinosis, ochronosis of the hip/knee joint
* slowly progressing hip/knee arthropathy in particular of tuberculosis aetiology
* hip/knee arthropathy due to diabetes mellitus
* Charcot's joint
* villous synovitis
* chondromatosis of the synovium
* patients with existing gastritis or existing ulcers or bleedings in the gastrointestinal tract or patients with history of gastrointestinal ulcers or gastrointestinal haemorrhage in the past 6 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 482 (Actual)
Dates: Start 2009-10; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Tolerability profile of Dexibuprofen Gebro 400 mg powder for oral suspension compared to Ibuprofen 400 mg in patients with painful osteoarthritis of the hip or knee | 14 days

SECONDARY OUTCOMES:
Overall efficacy of Dexibuprofen Gebro 400 mg powder for oral suspension compared to Ibuprofen 400 mg in patients suffering from different complaints due to painful osteoarthritis of the hip or knee | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Reinhold Hawel, MD, Principal Investigator — Rehabilitationszentrum, Bad Hofgastein
Locations (2):
- Austria (2):
  - Rehabzentrum für Erkrankungen des rheumat. Formenkreises, Bad Hofgastein, Salzburg
  - Rheuma Zentrum Favoriten, Vienna

REFERENCES:
- See also: Related Info — http://www.gebro.com